CLINICAL TRIAL: NCT07403448
Title: Effects of 9 Points Electrical Dry Needling on Pain, Range of Motion, Function and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Effects of 9 Points Electrical Dry Needling in Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0197
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Arthritis Osteoarthritis
Keywords: Arthritis, knee pain, Electrical dry needling, Grade 3 KOA, Functional limitations
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : 9 points electrical dry needling along with standard physical therapy (Experimental): 3 times per week for 6 weeks
  Interventions: Other: 9 points electrical dry needling; Other: Standard physical therapy
- active comparator: standard physical therapy (Active Comparator): 3 times per week for6 weeks
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: 9 points electrical dry needling — 9 points electrical dry needling, stainless steel dry needles of size 0.25 into 30mm will be used, inserted perpendicularly into popliteus, adductor magnus, tibialis anterior, quad tendon, vastus lateralis, medialis, medial & lateral infrapatellar sulcus, extensor digitorum longus.
  Arms: Experimental : 9 points electrical dry needling along with standard physical therapy
Other: Standard physical therapy — Standarized physical therapy: HOT pack for 5 min, hams & quads stretching for 30 sec & 6 reps, quads strengthening straight leg raise & leg press will be performed 15 reps & 3 sets, for hams seated leg curls & gluteal bridges will be performed 15 reps & 3 sets.
  MWM in weight bearing position: The glide will be applied in weight bearing, effected knee on stepper, the therapist will be exactly sitting in front of the patient & patient will be asked to place the limb up on the stepper one hand of the therapist has to be on the lateral side of the tibia and other hand on the medial side of the femur & now the patient will be asked to climb, therapist will apply medial & lateral pressure 10 reps & 3 sets.

SUMMARY:
The study will be conducted to compare effects of 9 points electrical dry needling along with standard physical therapy and standard physical therapy alone in knee osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* participants age group from 40-60 years
* Both male and female genders
* Knee osteoarthritis (OA) confirmed by radiographic evidence (Kellgren- Lawrence grade 3).
* Numerical Pain Rating Scale (NPRS) ≥ 4/10.
* Able to stand and bear weight on affected knee.
* WOMAC score > 25 moderate level of difficulty performing ADL
* Participant with restricted range of motion
* Pain while walking and ascending stairs
* Patients volunteered to participate in the study and signed informed consent

Exclusion Criteria:

* Mild to severe knee osteoarthritis (Kellgren-Lawrence grade 2 or 4).
* Recent knee surgery or injection (<6 months).
* Knee instability and ligamentous injury.
* Pregnancy and breastfeeding.
* Patient with needle phobia and with history of abnormal reaction to needles.
* Diagnosed psychological disorders
* Anticoagulant patient, tumors and hematomas.
* All acute emergencies and acute systematic fevers.
* Pacemakers and implantable cardioverter defibrillators

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | from enrollment to the end of 6 week
  Numeric Pain Rating Scale (NPRS) measures subjective pain intensity using an 11-point numeric scale (0-10) where 0 = "no pain" and 10 = "worst pain imaginable". Patients verbally or mark on a horizontal line the whole number best reflecting current pain severity, typically assessing "current pain," "worst pain," "least pain," or "average pain" over the prior 24 hours. Mild pain = 1-3, moderate pain = 4-6, severe pain = 7-10 guides clinical decision-making.
  changes in NPRS scale will be measured baseline and at the end of 6 week.
Goniometer measures joint range of motion (ROM) | from enrollment to the end of 6 week
  Goniometer: Precision instrument measuring joint range of motion (ROM) in degrees using protractor body with two arms (stationary and movable) aligned to anatomical bony landmarks spanning the joint axis.
  Primary Use: Quantifies active (AROM) and passive (PROM) joint excursion for objective baseline, progress tracking, and impairment rating. Universal goniometer most common; digital/smartphone apps offer improved reliability (ICC >0.9 vs 0.74-0.91 traditional).
  Reliability: Long-arm > short-arm (MSD 6° vs 10°); inter/intra-rater ICC 0.84-0.99 with standardized technique.
  changes in knee flexion and extension ROM will be measured baseline and at the end of 6 week.
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | from enrollment to the end of 6 week
  WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a validated, disease-specific patient-reported outcome measure for hip/knee osteoarthritis assessing pain (5 items, 0-20), stiffness (2 items, 0-8), and physical function (17 items, 0-68) over past 48 hours.
  Scoring: Likert 0-4 scale per item (0=None, 4=Extreme); higher total scores (0-96) indicate worse symptoms. MCID: 12% improvement (~9-12 points) represents clinically meaningful change.
  changes in WOMAC score will be measured baseline and at the end of 6 week.
EQ-5D 3L (QUALITY OF LIFE) | From enrollment to the end of 6 week
  EQ-5D-3L is developed by EuroQol groups is standardized instrument for measurement of health-related quality of life. it administers strong test-retest reliability for knee OA which of 0.73 to 0.91.
  Changes in EQ-5D 3L will be measured at baseline and at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Shakil ur Rehman, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Khalifa Bin Zayed Hospital, Quetta, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No